CLINICAL TRIAL: NCT01784276
Title: A PILOT AND FEASIBILITY STUDY OF ELECTRONIC SCREEN MEDIA TO REDUCE DENTAL FEAR AMONG CHILDREN WITH AUTISM SPECTRUM DISORDER
Brief Title: Dental Fear Among Children With Autism Spectrum Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Inyang Isong, MD, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-CRX10-09-0486-2
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2013-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Dental Fear
Keywords: Children; Autism Spectrum Disorders; Electronic Screen Media; Dental fear
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Children assigned to Group A (control group) received usual care and therefore had no intervention before or during the return visit.
- Video peer modeling (Experimental): Video peer modeling (at home, the child watched a DVD recording of a typically developing child undergoing a dental visit);
  Interventions: Behavioral: Video
- Video goggles or portable DVD only (Experimental): Video goggles/DVD (during the dental visit, the child watched their favorite movie using sunglass style video eyewear, or portable DVD player);
  Interventions: Behavioral: Video
- Video peer modeling plus video goggles (Experimental): Video peer modeling plus video goggles/DVD. At home, the child watched a DVD recording of a typically developing child undergoing a dental visit; During the dental visit, the child watched their favorite movie using sunglass style video eyewear, or portable DVD player.
  Interventions: Behavioral: Video

INTERVENTIONS:
Behavioral: Video — Video peer modeling: The video demonstrates various stages of the dental visit experience. Children assigned to intervention Groups B or D reviewed the video at least once, but as many times as possible before the follow up visit.
  Video goggles: This is a sunglass style video eyewear that contains two computer screens that can be used to watch 2 or 3D movies. Subjects randomized to Group C or D watched a 2D movie during the return visit, using the video goggles. Subjects who refused or were unable to wear the goggles watched the movie using a hand held portable DVD player.
  Arms: Video goggles or portable DVD only; Video peer modeling; Video peer modeling plus video goggles

SUMMARY:
Specific Aims Our study objective is to investigate if video peer modeling before the visit, plus immersive virtual reality during a preventive dental visit, reduces dental fear and uncooperative behaviors among children with ASD.

SPECIFIC AIM: To pilot and test the feasibility and effectiveness of video peer modeling and immersive virtual reality in reducing dental fear among children with autism undergoing preventive dental visits.

Methods: The investigators will enroll eighty (80) subjects aged 7-17 years with a known diagnosis of autism, who had a history of dental fear, per parental report.

Study hypotheses:

The primary hypotheses of interest are:

(i) The mean change in the Venham Anxiety Score (VAS) over the 4 month period in children with ASD who receive the video intervention (Group B) is different from the mean change in the VAS over the 4-month period in children with ASD in the control group.

(ii) The mean change in the VAS over the 4-month period in children with ASD who receive the immersive VR intervention (Group C) is different from the mean change in the VAS over the 4-month period in children with ASD in the control group.

(iii) The mean change in the VAS over the 4-month period in children with ASD who receive the video intervention plus the immersive VR intervention (Group D) is different from the mean change in the VAS over the 4-month period in children with ASD in the control group.

The secondary hypothesis is:

(i) The mean change in the Venham Behavior Score over the 4-month period in children with ASD in Group D is different from the mean change in the Venham Behavior Score over the 4-month period in children with ASD in Group B or C.

DETAILED DESCRIPTION:
Dental care is a significant unmet health care need for children with Autism Spectrum Disorders (ASD). Many children with ASD do not receive dental care because of fear associated with dental procedures; oftentimes they require general anesthesia for regular dental procedures, placing them at risk of associated complications. Many children with ASD have a strong preference for visual stimuli, particularly electronic screen media; this affinity has been utilized in their educational instruction.

Objective: To determine if an innovative strategy using two types of electronic screen media was feasible and beneficial in reducing fear and uncooperative behaviors in children with ASD undergoing dental visits.

Study procedures

For this randomized control study, we will randomize participants into one of 4 groups: a) control group (Group A); b) video peer modeling only group (Group B); c) immersive VR only group (Group C) and d) video peer modeling plus immersive VR group (Group D). All enrolled children will have a pre-visit in the dental clinic, where they will receive usual care and baseline values of all parameters will be obtained. Medical records of all study children will be flagged so that they are identified upon arrival by the RA. In the exam room, the dental assistant will measure their pulse rate using a pulse oximeter. The dentist and RA will complete the Venham Anxiety and Behavioral Scale during the dental procedure for all study children. All study subjects will be scheduled to return for a follow up preventive dental visit in 4-6 months, which is the usual practice at CHB, depending on the child's oral health status. Children assigned to intervention Groups B and D will be mailed a copy of a DVD of the pre-recorded peer modeled visit 4 weeks before the scheduled return for the preventive dental visit. The parents will be asked to review the video with their child to orient them to all stages of the dental visit. In addition, children assigned to Group C and D will be given a virtual reality headset to watch movies or images during the dental visit. Children assigned to Group A (control group) will receive neither the DVD nor VR headset during the visit. We will repeat all measurements during the return visit for all study children.

Participant randomization: Once we identify the entire sample of eligible subjects, we will generate a list of subjects that have enrolled for the study. With the assistance of the statistician, we will do a random allocation of each subject to Group A, B, C or D.

Sample size calculation:

In order to have an 80% chance of detecting a difference of 1 unit in either the mean change in the Venham anxiety score (VAS) over the 4-month period in children with ASD assigned to Group B, C or D, with the mean change in the VAS over the 4-month period in children with ASD in Group A, allowing for a 20% dropout rate, a total sample size of 80 children will be required. Subjects are being allocated equally between the 4 groups and each group will be randomly assigned 20 subjects. Data Analyses: After obtaining values of the Venham Anxiety and Behavior Scores for each group at baseline and 4 month period, the change in score will be calculated for each subject and a mean change in score and standard deviation generated for each group. WE will use a two-sided t-test to test each of these hypotheses. Bonferroni adjustments will be used to account for the multiple comparisons being carried out. The association of important covariates, such as the level of cognitive functioning, IQ, age, gender and number of hours of ABA received with the change in VAS will be modeled using linear regression analyses, with the outcome variable being the mean change in score for each subject. (A separate model will be fit for each outcome variable). Further analyses will include examining the association of pulse rate (a continuous outcome measure) with the covariates listed above. All analyses will be conducted by the study statistician and PI.

Data Management Methods The RA will collect and manage all study data. We will enter personal information of study subjects obtained at enrollment in the study database. All subjects will be assigned codes which will be used throughout the study. No subject identifying personal information will be used to make up the study code for a specific patient. The link between the study-ID and medical record number will be kept in a locked/double password protected file. The Dr Isong and the RA will be the only ones who know the key/passwords.

Data and Safety Monitoring Plan Every 6 months, all study data and protocols will be reviewed by the RA and PI to ensure that they confirm to written stipulations. Any missing data will be noted and collected.

To prevent disclosure, information about participation and the results of the research will not be placed in the medical record. Study data will be coded and the key to the code kept in a separate locked file. All research data will be entered into a database. No names are entered into this database, only the codes assigned to the research record. All results will remain confidential. Only anonymized data will be shared among collaborators.

Safety monitoring Risks associated with this study are expected to be minimal. Any report of risk or discomfort as a result of the study (please see below) experienced by study subjects will be documented and appropriate treatment and referrals will be provided. Subjects will be informed that they can dis-enroll from the study at any time if they experience any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 7-17 years with a known diagnosis of autism, who had a history of dental fear, per parental report.

Exclusion Criteria:

* children with motor handicaps (e.g. cerebral palsy), and sensory, vision and hearing impairments (as these would have limited their ability to utilize intervention materials);
* children with parents who did not speak English or Spanish; and
* children who presented to clinic without their legal guardian.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Anxiety | 6 month
  Primary outcome:
  Anxiety: To assess the subject's level of anxiety, we will use the Venham Anxiety Rating Scale which assigns numerical values to the child's observable behaviors. It consists of 5 behaviorally defined categories that range from 0-5, and higher scores indicate greater levels of anxiety.(ref) The treating dentist and RA will use the Venham Scale to indicate their perception of level of anxiety experienced by the participant during the dental procedure.

SECONDARY OUTCOMES:
Uncooperative behavior | 6 month
  Behavior: To assess the subject's behavior during the dental visit, we will use the Venham Behavior Rating Scale.(ref) The Behavior Scale also consists of 5 behaviorally defined categories that range from 0-5, and higher scores indicate greater levels of uncooperative behavior.(ref) The Venham Anxiety and Behavior Rating Scales have been used extensively in behavior research to assess the level of anxiety and behavior of children in dental settings.(ref) The RA and treating dentist will rate te child's behavior once during the dental visit. The PI will train the dentist and RA on procedures to administer the Venham Anxiety and Behavior Rating Scale during the dental visit and will assess inter-rater reliability.

OTHER OUTCOMES:
Pulse rate | 6 months
  Physiological arousal: We will obtain the child's pulse rate as an objective measure of physiological arounsal during the dental procedure. The dental assistant will use a pulse oximeter to measure the pulse rate at three time points: - after the child is brought into the examination room, about 15 minutes into the dental procedure and about 5 minutes after the dental procedure is completed.

CONTACTS AND LOCATIONS:
Overall Officials: INYANG ISONG, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children'S Hospital, Boston, Massachusetts, United States